CLINICAL TRIAL: NCT01103713
Title: An Open Label, Non-comparative Study To Evaluate Parasitological Clearance Rates And Pharmacokinetics Of Azithromycin And Chloroquine Following Administration Of A Fixed Dose Combination Of Azithromycin And Chloroquine (Azcq) In Asymptomatic Pregnant Women With Plasmodium Falciparum Parasitemia In Sub-saharan Africa
Brief Title: Evaluate Parasitological Clearance Rates And Pharmacokinetics Of The Combination Of Azithromycin And Chloroquine In Asymptomatic Pregnant Women With Falciparum Parasitemia In Africa
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0661201
Record Dates: First submitted 2010-04-07; First posted 2010-04-15 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Asymptomatic Parasitemia In Pregnancy
Keywords: P. falciparum malaria; asymptomatic parasitemia; parasitological clearance; Intermittent Preventive Treatment of Falciparum Malaria in Pregnant Women (IPTp)
MeSH Terms: interventions — Azithromycin; Chloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AZCQ (Experimental): Azithromycin/Chloroquine
  Interventions: Drug: Azithromycin plus chloroquine

INTERVENTIONS:
Drug: Azithromycin plus chloroquine — Study drug is a fixed dose tablet of AZCQ containing 250 mg AZ and 155 mg CQ base. All subjects will be administered a 3 day course of AZCQ IPTp regimen: a single dose of 1000 mg AZ/620 mg CQ base (4 fixed dose combination tablets of AZCQ: 250mg/155mg) administered per os (PO, orally) once daily for 3 days (Days 0, 1, 2).
  Other Names: Zithromax; Aralen

SUMMARY:
The study will be conducted in asymptomatic pregnant women with P. falciparum parasitemia. The subjects will be given 3 day dosing regiment of the fixed-dose combination of Azithromycin and Chloroquine. Parasitological clearance rate with polymerase chain reaction data will be evaluated on Day 28 as primary endpoint.

DETAILED DESCRIPTION:
After interim analysis of efficacy data by an External Data Monitoring Committee, this study was terminated. Investigators were notified on 22 Aug 2013. There were no safety concerns that led to this termination.

ELIGIBILITY:
Inclusion Criteria:

* Primigravidae and secundigravidae pregnant women at >=14 and <=30 weeks of gestational age (confirmed by ultrasound examination).
* Evidence of asymptomatic parasitemia with Plasmodium falciparum monoinfection (confirmed by microscopy) with parasite counts in the range of 80 100,000/uL on thick blood smears.
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative if a subject is <18 years of age) has been informed of all pertinent aspects of the study and that all questions by the subject have been sufficiently answered. Assent will be obtained from subjects <18 years of age.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Age <16 years old or >35 years old.
* Multiple gestations (more than one fetus) as per the ultrasound results at screening.
* Clinical symptoms of malaria.
* Hemoglobin <8 g/dL (measured at baseline).
* Any condition requiring hospitalization or evidence of severe concomitant infection at time of presentation.
* Use of antimalarial drugs in previous 4 weeks.
* History of convulsions, hypertension, diabetes or any other chronic illness that may adversely affect fetal growth and viability.
* Known allergy to the study drugs (AZ, CQ, and SP) or to any macrolides or sulphonamides.
* Requirement to use medication during the study that might interfere with the evaluation of the study drug of AZ or CQ or is contra indicated during pregnancy per package inserts.
* Severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
* Evidence of current obstetric complications that may adversely impact the pregnancy and/or fetal outcomes, including presence of congenital anomalies, placenta previa or abruption.
* Known severe sickle cell (SS) disease or sickle hemoglobin C (SC) anemia.
* Known family history of prolonged QT syndrome, serious ventricular arrhythmia, or sudden cardiac death.

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 168 (Actual)
Dates: Start 2011-03; Primary Completion 2013-06 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- Benin (2):
  - Centre de Sante d'AHOUANSORI -AGUE, Cotonou
  - Hôpital Bethesda, Cotonou
- Siaya District Hospital, Siaya, Kenya
- Zomba Central Hospital, Zomba, Malawi
- Tanzania (2):
  - Teule Hospital, Muheza, Tanga
  - National Institute for Medical Research (Mwanza Centre)/ Nyamagana District Hospital, Mwanza
- Mulanda Health Centre IV, Kampala, Uganda

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661201&StudyName=Evaluate%20Parasitological%20Clearance%20Rates%20And%20Pharmacokinetics%20Of%20The%20Combination%20Of%20Azithromycin%20And%20Chloroquine%20In%20Asymptomatic%20Pregnant%20Wome

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 5 active sites in 5 countries: Benin (site 1012), Kenya (site 1004), Malawi (site 1015), Tanzania (site 1008), and Uganda (site 1013). The enrollment of the first participant took place on 07 March 2011 and the last participant last visit was on 25 October 2013.
Pre-assignment Details: A total of 404 participants were screened and 168 participants were assigned to study drug, enrolled and treated. Of the 168 participants, two participants were excluded from the pharmacokinetic (PK) analysis, modified intent-to-treat (MITT), intent-to-treat (ITT) and per protocol (PP) populations due to informed consent protocol deviations.
Groups:
- Azithromycin (AZ)/Chloroquine (CQ): Study drug AZCQ is a fixed dose combination tablet of AZ and CQ containing 250 mg AZ and 155 mg CQ base. The dosing regimen evaluated in this study consisted of four AZCQ tablets (a total of 1000 mg AZ/620 mg CQ base), given orally once daily for 3 days (Days 0, 1, 2).
Period: Overall Study
Arm/Group | Azithromycin (AZ)/Chloroquine (CQ)
Started | 168
Completed | 155
Not Completed | 13
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 8
Not completed — Study terminated by sponsor | 2
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Azithromycin (AZ)/Chloroquine (CQ)
Number analyzed (Participants) | 168
Age, Customized [Number; unit: Participants]
  <16 years | 0
  16-17 years | 41
  18-25 years | 125
  26-30 years | 1
  31-35 years | 1
  >35 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Parasitologic Response (Polymerase Chain Reaction (PCR) Corrected) at Day 28 Post First Dose of Study Medication
Description: The proportion of participants with parasitological response was estimated from the Kaplan Meier curve based on the time to the first occurrence of parasitological failure (PCR corrected). A participant will be a parasitological responder if she has a zero parasite count on the Day 7 visit without subsequent recurrence (PCR corrected) through the day of consideration, otherwise she is a parasitological failure.
Time Frame: Day 28
Population: MITT population was used. MITT is a subset of the ITT population who had Plasmodium falciparum monoinfection (confirmed by microscopy) parasite count in the range of 80-100,000/microlitre on their baseline blood smear. Two participants were excluded because they had protocol deviations regarding the informed consent process.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Azithromycin (AZ)/Chloroquine (CQ)
Number analyzed (Participants) | 163
Percentage of participants | 99.35 [97.76 to 100.00]

2. Primary Outcome: Percentage of Participants With Parasitologic Response (PCR Corrected) at Day 28 Post First Dose of Study Medication
Description: as for outcome 1
Time Frame: Day 28
Population: PP population was used. PP is a subset of MITT population who had received all 3 days of study medication. Two participants were excluded because they had protocol deviations regarding the informed consent process.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Azithromycin (AZ)/Chloroquine (CQ)
Number analyzed (Participants) | 158
Percentage of participants | 99.35 [97.76 to 100.00]

3. Secondary Outcome: Percentage of Participants With Parasitologic Response (PCR Corrected) at Days 7, 14, 21, 35, and 42 Post First Dose of Study Medication
Description: as for outcome 1
Time Frame: Days 7, 14, 21, 35, and 42
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Azithromycin/Chloroquine (AZCQ): This is an open label, single arm study conducted in pregnant women during their second and third trimesters of pregnancy. Study drug AZCQ is a fixed dose combination tablet of AZ and CQ containing 250 mg AZ and 155 mg CQ base. The dosing regimen evaluated in this study consisted of four AZCQ tablets (a total of 1000 mg AZ/620 mg CQ base), given orally once daily for 3 days (Days 0, 1, 2).
Arm/Group | Azithromycin/Chloroquine (AZCQ)
Number analyzed (Participants) | 163
Percentage of participants
  Day 7 (n=156) | 100 [97.66 to 100.00]
  Day 14 (n=154) | 100 [97.63 to 100.00]
  Day 21 (n=154) | 100 [97.63 to 100.00]
  Day 35 (n=148) | 96.65 [93.42 to 99.87]
  Day 42 (n=138) | 95.19 [91.35 to 99.03]

4. Secondary Outcome: Percentage of Participants With Parasitologic Response (PCR Corrected) at Days 7, 14, 21, 35, and 42 , Post First Dose of Study Medication
Description: as for outcome 1
Time Frame: Days 7, 14, 21, 35, and 42
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Azithromycin (AZ)/Chloroquine (CQ)
Number analyzed (Participants) | 158
Percentage of participants
  Day 7 (n=156) | 100.00 [97.66 to 100.00]
  Day 14 (n=154) | 100.00 [97.63 to 100.00]
  Day 21 (n=154) | 100.00 [97.63 to 100.00]
  Day 35 (n=148) | 96.65 [93.42 to 99.87]
  Day 42 (n=138) | 95.19 [91.35 to 99.03]

5. Secondary Outcome: Percentage of Participants With Parasitologic Response (PCR Corrected) at Days 7, 14, 21, 28, 35, and 42 Post First Dose of Study Medication
Description: as for outcome 1
Time Frame: Days 7, 14, 21, 28, 35, and 42
Population: ITT population was used. ITT is defined as all participants who received at least one dose of study medication and who had a baseline blood smear positive for Plasmodium falciparum monoinfection, asexual parasitemia. Two participants were excluded because they had protocol deviations regarding the informed consent process.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Azithromycin (AZ)/Chloroquine (CQ)
Number analyzed (Participants) | 165
Percentage of participants
  Day 7 (n=158) | 100.00 [97.69 to 100.00]
  Day 14 (n=156) | 100.00 [97.66 to 100.00]
  Day 21 (n=156) | 100.00 [97.66 to 100.00]
  Day 28 (n=156) | 99.36 [97.79 to 100.00]
  Day 35 (n=150) | 96.69 [93.51 to 99.88]
  Day 42 (n=140) | 95.26 [91.47 to 99.05]

6. Secondary Outcome: Percentage of Participants With Parasitologic Response (PCR Uncorrected) at Days 7, 14, 21, 28, 35, and 42 Post First Dose of Study Medication
Description: The proportion of participants with parasitological response was estimated from the Kaplan Meier curve based on the time to the first occurrence of parasitological failure (PCR uncorrected). A participant will be a parasitological responder if she has a zero parasite count on the Day 7 visit without subsequent recurrence (PCR uncorrected) through the day of consideration, otherwise she is a parasitological failure.
Time Frame: Days 7, 14, 21, 28, 35, and 42
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Azithromycin (AZ)/Chloroquine (CQ)
Number analyzed (Participants) | 163
Percentage of participants
  Day 7 (n=156) | 100.00 [97.66 to 100.00]
  Day 14 (n=154) | 100.00 [97.63 to 100.00]
  Day 21 (n=154) | 100.00 [97.63 to 100.00]
  Day 28 (n=154) | 95.45 [91.84 to 99.07]
  Day 35 (n=154) | 87.66 [82.14 to 93.18]
  Day 42 (n=152) | 78.43 [71.59 to 85.28]

7. Secondary Outcome: Percentage of Participants With Parasitologic Response (PCR Uncorrected) at Days 7, 14, 21, 28, 35, and 42 Post First Dose of Study Medication
Description: as for outcome 6
Time Frame: Days 7, 14, 21, 28, 35, and 42
Population: PP population was used. PP is a subset of MITT population who received all 3 days of study medication. Two participants were excluded because they had protocol deviations regarding the informed consent process.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Azithromycin (AZ)/Chloroquine (CQ)
Number analyzed (Participants) | 158
Percentage of participants
  Day 7 (n=156) | 100.00 [97.66 to 100.00]
  Day 14 (n=154) | 100.00 [97.63 to 100.00]
  Day 21 (n=154) | 100.00 [97.63 to 100.00]
  Day 28 (n=154) | 95.45 [91.84 to 99.07]
  Day 35 (n=154) | 87.66 [82.14 to 93.18]
  Day 42 (n=152) | 78.43 [71.59 to 85.28]

8. Secondary Outcome: Percentage of Participants With Parasitologic Response (PCR Uncorrected) at Days 7, 14, 21, 28, 35, and 42 Post First Dose of Study Medication
Description: as for outcome 6
Time Frame: Days 7, 14, 21, 28, 35, and 42
Population: ITT population was used. ITT is defined as all participants who received at least one dose of study medication and had a baseline blood smear positive for Plasmodium falciparum monoinfection, asexual parasitemia. Two participants were excluded because they had protocol deviations regarding the informed consent process.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Azithromycin (AZ)/Chloroquine (CQ)
Number analyzed (Participants) | 165
Percentage of participants
  Day 7 (n=158) | 100.00 [97.69 to 100.00]
  Day 14 (n=156) | 100.00 [97.66 to 100.00]
  Day 21 (n=156) | 100.00 [97.66 to 100.00]
  Day 28 (n=156) | 95.51 [91.94 to 99.08]
  Day 35 (n=156) | 87.82 [82.37 to 93.27]
  Day 42 (n=154) | 78.71 [71.94 to 85.48]

9. Secondary Outcome: Number of Asexual P. Falciparum Per Microliter of Blood at Days 7, 14, 21, 28, 35, and 42 Post First Dose of Study Medication
Description: Parasite counts (actual counts per microliter of blood) was measured at various time points.
Time Frame: Days 7, 14, 21, 28, 35, and 42
Population: as for outcome 8
Measure: Mean (Standard Error); unit: Parasite count per microliter
Arm/Group | Azithromycin (AZ)/Chloroquine (CQ)
Number analyzed (Participants) | 165
Parasite count per microliter
  Day 7 (n=155) | 0.00 (0.00)
  Day 14 (n=154) | 0.00 (0.00)
  Day 21 (n=156) | 0.00 (0.00)
  Day 28 (n=156) | 216.91 (110.04)
  Day 35 (n=156) | 555.36 (246.77)
  Day 42 (n=155) | 907.88 (470.82)

10. Secondary Outcome: Number of Asexual P. Falciparum Per Microliter of Blood at Days 7, 14, 21, 28, 35, and 42 Post First Dose of Study Medication
Description: Parasite counts (actual counts per microliter of blood) was measured at various time points.
Time Frame: Days 7, 14, 21, 28, 35, and 42
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Parasite count per microliter
Arm/Group | Azithromycin (AZ)/Chloroquine (CQ)
Number analyzed (Participants) | 163
Parasite count per microliter
  Day 7 (n=153) | 0.00 (0.00)
  Day 14 (n=152) | 0.00 (0.00)
  Day 21 (n=154) | 0.00 (0.00)
  Day 28 (n=154) | 219.73 (111.46)
  Day 35 (n=154) | 562.57 (249.94)
  Day 42 (n=153) | 919.75 (476.92)

11. Secondary Outcome: Number of Asexual P. Falciparum Per Microliter of Blood at Days 7, 14, 21, 28, 35, and 42 Post First Dose of Study Medication
Description: Parasite counts (actual counts per microliter of blood) was measured at various time points.
Time Frame: Days 7, 14, 21, 28, 35, and 42
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Parasite count per microliter
Arm/Group | Azithromycin (AZ)/Chloroquine (CQ)
Number analyzed (Participants) | 158
Parasite count per microliter
  Day 7 (n=153) | 0.00 (0.00)
  Day 14 (n=152) | 0.00 (0.00)
  Day 21 (n=154) | 0.00 (0.00)
  Day 28 (n=154) | 219.73 (111.46)
  Day 35 (n=154) | 562.57 (249.94)
  Day 42 (n=153) | 919.75 (476.92)

12. Other Pre Specified Outcome: Summary of Pregnancy Outcome: Location of Delivery
Description: All participants were followed up for exposure-in-utero (EIU) safety assessments following delivery or termination of pregnancy.
Time Frame: Following delivery or pregnancy termination
Population: The safety analysis set consists of participants who received at least one dose of study medication. Data was available for 160 participants only.
Measure: Number; unit: Participants
Arm/Group | Azithromycin (AZ)/Chloroquine (CQ)
Number analyzed (Participants) | 160
Participants
  Medical facility | 130
  Home | 27
  Other (Not specified) | 3

13. Other Pre Specified Outcome: Summary of Pregnancy Outcome: Mode of Delivery
Description: All participants were followed up for EIU safety assessments following delivery or termination of pregnancy.
Time Frame: Following delivery or pregnancy termination
Population: as for outcome 12
Measure: Number; unit: Participants
Arm/Group | Azithromycin (AZ)/Chloroquine (CQ)
Number analyzed (Participants) | 160
Participants
  Vaginal | 145
  Cesarean section | 15

14. Other Pre Specified Outcome: Summary of Pregnancy Outcome: Delivery Assisted by Trained Obstetric Personnel?
Description: All participants were followed up for EIU safety assessments following delivery or termination of pregnancy.
Time Frame: Following delivery or pregnancy termination
Population: The safety analysis set consists of participants who received at least one dose of study medication. Data was available for 159 participants only.
Measure: Number; unit: Participants
Arm/Group | Azithromycin (AZ)/Chloroquine (CQ)
Number analyzed (Participants) | 159
Participants
  Yes | 132
  No | 27

15. Other Pre Specified Outcome: Summary of Pregnancy Outcome: Labor Induced?
Description: All participants were followed up for EIU safety assessments following delivery or termination of pregnancy.
Time Frame: Following delivery or pregnancy termination
Population: The safety analysis set consists of participants who received at least one dose of study medication. Data was available for 158 participants only.
Measure: Number; unit: Participants
Arm/Group | Azithromycin (AZ)/Chloroquine (CQ)
Number analyzed (Participants) | 158
Participants
  Yes | 3
  No | 155

16. Other Pre Specified Outcome: Summary of Pregnancy Outcome: Complications During Delivery?
Description: All participants were followed up for EIU safety assessments following delivery or termination of pregnancy.
Time Frame: Following delivery or pregnancy termination
Population: as for outcome 14
Measure: Number; unit: Participants
Arm/Group | Azithromycin (AZ)/Chloroquine (CQ)
Number analyzed (Participants) | 159
Participants
  Yes | 42
  No | 117

17. Other Pre Specified Outcome: Summary of Pregnancy Outcome: Outcome of Birth
Description: All participants were followed up for EIU safety assessments following delivery or termination of pregnancy.
Time Frame: Following delivery or pregnancy termination
Population: as for outcome 12
Measure: Number; unit: Participants
Arm/Group | Azithromycin (AZ)/Chloroquine (CQ)
Number analyzed (Participants) | 160
Participants
  Full term live birth | 151
  Premature birth | 6
  Stillbirth | 3
  Spontaneous abortion | 0
  Induced/elective abortion | 0

18. Other Pre Specified Outcome: Incidence of Fever Based on Oral Temperature
Description: Oral temp was taken by the fieldworker through Day 42.
Time Frame: Baseline, Days 1, 2, 7, 14, 21, 28, 35, and 42
Population: ITT is defined as all participants who received at least one dose of study medication and who had a baseline blood smear positive for Plasmodium falciparum monoinfection, asexual parasitemia. Two participants were excluded because they had protocol deviations regarding the informed consent process.
Measure: Number; unit: Participants
Arm/Group | Azithromycin (AZ)/Chloroquine (CQ)
Number analyzed (Participants) | 168
Participants
  Baseline (n=165) | 0
  Day 1 (n=161) | 0
  Day 2 (n=160) | 0
  Day 7 (n=156) | 0
  Day 14 (n=155) | 0
  Day 21 (n=155) | 0
  Day 28 (n=156) | 0
  Day 35 (n=156) | 0
  Day 42 (n=155) | 4

19. Other Pre Specified Outcome: Summary of Hemoglobin Concentration: Abnormal Hemoglobin Level
Description: Abnormal hemoglobin level on Day 42 was measured. The hemoglobin levels were measured with HemoCueTM, via finger stick or peripheral blood collection. The reference range was 10-16g/dL. Any value <0.8 times lower limit of normal was considered clinically significant.
Time Frame: Day 42
Population: The safety analysis set consists of participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Azithromycin (AZ)/Chloroquine (CQ)
Number analyzed (Participants) | 168
Participants | 1

20. Other Pre Specified Outcome: Summary of Serum Azithromycin Concentration Versus Time
Description: AZ concentrations in the serum was determined at specified time points as PK endpoints
Time Frame: Planned time: 0 (Day 0), 48 (Day 2), 50 (Day 2), 56 (Day 2), 168 (Day 7), and 336 (Day 14) hours post the first dose. Note: Assuming "hour not specified" as 0 hours on Day 7 and Day 14 for planned time post first dose calculation.
Population: Analyses population included all participants who received at least one dose of study medication and had at least one blood sample collected for PK analysis.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Azithromycin (AZ)/Chloroquine (CQ)
Number analyzed (Participants) | 166
ng/ml
  Hour 0 (Day 0) (n=161) | NA (NA) — Summary statistics have been calculated by setting concentration values below the low limit of quantification to zero.
  Hour 48 (Day 2) (n=158) | 194.145 (63.76829)
  Hour 50 (Day 2) (n=147) | 994.463 (552.23738)
  Hour 56 (Day 2) (n=159) | 707.682 (326.72379)
  Hour 168 (Day 7) (n=155) | 54.444 (24.34615)
  Hour 336 (Day 14) (n=153) | 20.307 (31.57879)

21. Other Pre Specified Outcome: Summary of Plasma Chloroquine Concentration Versus Time
Description: CQ concentrations in the plasma were determined at specified time points as PK endpoints
Time Frame: Planned time: 0 (Day 0), 48 (Day 2), 50 (Day 2), 56 (Day 2), 168 (Day 7), 336 (Day 14), 504 (Day 21) and 672 (Day 28) post first dose. Note: Assuming "hour not specified" as 0 hours on Days 7, 14, 21 and 28 for planned time post first dose calculation.
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Azithromycin (AZ)/Chloroquine (CQ)
Number analyzed (Participants) | 166
ng/ml
  Hour 0 (Day 0) (n=160) | NA (NA) — Summary statistics have been calculated by setting concentration values below the low limit of quantification to zero.
  Hour 48 (Day 2) (n=158) | 305.827 (129.02771)
  Hour 50 (Day 2) (n=147) | 621.134 (329.92731)
  Hour 56 (Day 2) (n=159) | 640.679 (297.97628)
  Hour 168 (Day 7) (n=155) | 129.835 (92.19161)
  Hour 336 (Day 14) (n=154) | 43.119 (44.97312)
  Hour 504 (Day 21) (n=156) | 22.382 (46.83029)
  Hour 672 (Day 28) (n=156) | 12.721 (29.05380)

22. Other Pre Specified Outcome: Summary of Plasma Desethylchloroquine Concentration Versus Time
Description: CQ concentrations in the plasma were determined at specified time points as PK endpoints
Time Frame: as for outcome 21
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Azithromycin (AZ)/Chloroquine (CQ)
Number analyzed (Participants) | 166
ng/ml
  Hour 0 (Day 0) (n=158) | NA (NA) — Summary statistics have been calculated by setting concentration values below the low limit of quantification to zero.
  Hour 48 (Day 2) (n=158) | 183.622 (118.86488)
  Hour 50 (Day 2) (n=147) | 220.424 (130.48349)
  Hour 56 (Day 2) (n=159) | 241.831 (137.88581)
  Hour 168 (Day 7) (n=155) | 144.088 (123.66303)
  Hour 336 (Day 14) (n=154) | 55.513 (54.78967)
  Hour 504 (Day 21) (n=156) | 29.825 (32.41800)
  Hour 672 (Day 28) (n=156) | 19.439 (19.52079)

ADVERSE EVENTS:
Time Frame: Day 42 follow-up visit for treatment emergent AEs for mothers and 14 days post delivery for neonates
Description: No treatment emergent serious adverse events (SAEs) were observed in mothers. Events related to neonatal malformation/anomalies, premature delivery, low birth weight neonates, developmental assessment, kernicterus, or any other neonatal illness, hospitalization, drug therapy etc, were recorded and presented under the "familial status = neonates"
Groups:
- Azithromycin/Chloroquine (Familial Status = Neonate): AZCQ (Familial Status = Neonate)
- Azithromycin/Chloroquine (Familial Status = Mother): ACZQ (Familial Status = Mother)
Arm/Group | Azithromycin/Chloroquine (Familial Status = Neonate) | Azithromycin/Chloroquine (Familial Status = Mother)
Serious Adverse Events (participants affected / at risk) | 9/157 | 0/168
Other Adverse Events (participants affected / at risk) | 20/157 | 92/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Azithromycin/Chloroquine (Familial Status = Neonate) (N=157) | Azithromycin/Chloroquine (Familial Status = Mother) (N=168)
Hypospadias (Congenital, familial and genetic disorders) | 1 | 0/0
Polydactyly (Congenital, familial and genetic disorders) | 1 | 0/0
Sudden infant death syndrome (General disorders) | 1 | 0/0
Sepsis neonatal (Infections and infestations) | 1 | 0/0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 1 | 0/0
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 4 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azithromycin/Chloroquine (Familial Status = Neonate) (N=157) | Azithromycin/Chloroquine (Familial Status = Mother) (N=168)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 3
Food poisoning (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 6
Vomiting (Gastrointestinal disorders) | 0 | 35
Asthenia (General disorders) | 0 | 3
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 7
Pain (General disorders) | 0 | 1
Infection parasitic (Infections and infestations) | 0 | 12
Malaria (Infections and infestations) | 0 | 8
Trichomoniasis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 7
Urinary tract infection (Infections and infestations) | 0 | 4
Vulvovaginal candidiasis (Infections and infestations) | 0 | 4
White blood cells urine positive (Investigations) | 0 | 1 — Familial Status= Mother
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 33
Headache (Nervous system disorders) | 0 | 10
False labour (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 13
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 9
Macrosomia (General disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Neonatal infection (Infections and infestations) | 1 | 0
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 8 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 6 | 0
Umbilical cord around neck (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.